CLINICAL TRIAL: NCT02519088
Title: A New Approach to a Personalized Patient Blood Management Program in Total Hip Arthroplasty
Brief Title: A New Approach to a Personalized Patient Blood Management Program (pPBM) in Total Hip Arthroplasty (THA)
Status: Completed | Type: Observational
Sponsor: Krankenhaus der Barmherzigen Brüder Trier (Other)
Responsible Party: Principal Investigator, Ion-Andrei Popescu, MD, Ion-Andrei Popescu, MD, Krankenhaus der Barmherzigen Brüder Trier
Other Study IDs: KrankenhausBBT
Record Dates: First submitted 2015-08-03; First posted 2015-08-10 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Postoperative Anemia
Keywords: Homologous Blood Transfusion; Total Hip Replacement; Patient Blood Management

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study evaluates the patient related risk and predictive factors concerning perioperative homologous blood cell transfusion (erythrocyte concentrate ) in THA patients in one EndoCert max-certified orthopedic hospital in Germany.

A patient oriented preoperative decision-making algorithm (a personalised Patient Blood Management or pPBM App) will be developed as a new patient-safety blood-sparing strategy.

The aim is to increase the patient safety by using the pPBM App and to reach a more efficient management of resources.

DETAILED DESCRIPTION:
Retrospective audit of 470 consecutive primary THA in 2013 and 2014

ELIGIBILITY:
Inclusion Criteria:

* primary THA on patients with coxarthrosis

Exclusion Criteria:

* any kind of old or acute fractures about the basin and hip
* combined surgery, like first extracting a femur nail and than undergoing THA
* any other kind of combined or simultaneous surgery
* any kind of coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who electively underwent primary THA in 2013 and 2014
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Events and circumstances of Homologous Blood Transfusion (erythrocyte concentrate transfusion) | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Multivariate analysis of predictive variables like age, sex, BMI, hip and belly circumference, chronic kidney disease, chronic cardio-vascular disease, chronic inflammatory disease, diabetes mellitus, cancer, ASA Score, cemented, hybrid or not cemented prosthesis, surgery duration, medication and hemoglobin level before surgery

SECONDARY OUTCOMES:
pPBM Computer Simulation | participants will be followed for the duration of hospital stay, an expected average of 10 days
  Introducing the pPBM App as a safe blood-sparing strategy

CONTACTS AND LOCATIONS:
Overall Officials: Ion-Andrei Popescu, MD, Principal Investigator — Krankenhaus der Barmherzigen Brüder Trier
Locations (1):
- Krankenhaus der Barmherzigen Brüder Trier, Trier, Rhineland-Palatinate, Germany